CLINICAL TRIAL: NCT06360900
Title: Synergistic Gut-brain Axis Modulation Via Vagal Stimulation and Support Therapy in Functional Dyspepsia
Acronym: CONVERGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Roberta Sclocco, Assistant Professor, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024P000849; R01DK136243 (NIH)
Record Dates: First submitted 2024-04-03; First posted 2024-04-11 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Functional Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sensory device + Skills Building (Experimental)
  Interventions: Device: Sensory device; Behavioral: Skills Building
- Sensory device + Health Education (Active Comparator)
  Interventions: Device: Sensory device; Behavioral: Health Education
- Subsensory device + Skills Building (Active Comparator)
  Interventions: Behavioral: Skills Building; Device: Subsensory device
- Subsensory device + Health Education (Sham Comparator)
  Interventions: Behavioral: Health Education; Device: Subsensory device

INTERVENTIONS:
Device: Sensory device — Sensory vagal nerve stimulation
  Arms: Sensory device + Health Education; Sensory device + Skills Building
Behavioral: Skills Building — Skills Building behavioral therapy
  Arms: Sensory device + Skills Building; Subsensory device + Skills Building
Behavioral: Health Education — Education of FD condition
  Arms: Sensory device + Health Education; Subsensory device + Health Education
Device: Subsensory device — Subsensory vagal nerve stimulation
  Arms: Subsensory device + Health Education; Subsensory device + Skills Building

SUMMARY:
The study aims at evaluating physiological and patient-reported outcomes for a dual intervention approach including a stimulation device and support therapy in patients with functional dyspepsia.

ELIGIBILITY:
Inclusion Criteria:

Age 18-65 years old (inclusive)

* Ability to give written consent and participate in behavioral intervention in English
* Willingness to attend weekly treatment sessions over live video, daily self-administered transcutaneous auricular vagus nerve stimulation (taVNS) sessions, and engage in homework during treatment
* Avoidance of alcohol, nicotine, and caffeine for 24 hours prior to study session
* Diagnosis according to the Rome IV criteria for both epigastric pain syndrome and postprandial distress syndrome subtypes
* Stable medical treatment for functional dyspepsia (FD) during 1 month before the study and during the study period

Exclusion Criteria:

* Previous receipt of cognitive behavioral therapy (CBT) for gastrointestinal symptoms
* Enteral or parenteral feeding
* Previous gastrointestinal surgery, electrolyte disturbances, kidney dysfunction, renal insufficiency, or iron overload disorders
* Estimated Glomerular Filtration Rate (eGFR) < 60
* Medications that affect gastrointestinal motility in addition to medications or products containing tetrahydrocannabinol (THC) will be stopped at least 7 days prior to the start of the study and for the duration of the study. However, anti-depressants (SSRI's, TCA's) may be allowed in order to reduce the risk of worsening neuropsychiatric disease, though it will be up to the study team and the Principal Investigator whether subjects on anti-depressants will be able to participate in the study
* Intellectual disability by history
* Diabetes, mitochondrial disease, severe autonomic dysfunction, and small fiber polyneuropathy
* No active clinical acupuncture therapy
* Illicit drugs or opioid usage
* History of arrhythmias
* Current pregnancy/breastfeeding
* Contraindications for magnetic resonance imaging (MRI) (implanted ferromagnetic objects, claustrophobia)
* Weight > 450 lbs. (limit of the MRI table)
* Allergy to pineapple (used in the test meal during MRI)
* Any other condition interfering with study requirements, according to the Investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Visceral Sensitivity Index (VSI) | 8 weeks (post-treatment)
  GI-related anxiety; score ranging from score ranging from 0 to 75, with higher scores indicating worse outcomes

SECONDARY OUTCOMES:
Gastric peristaltic velocity | 8 weeks (post-treatment)
  MRI-derived gastric motility outcome
Nepean Dyspepsia Index (NDI) | 8 weeks (post-treatment)
  FD symptoms severity; score ranging from 0 to 100, with higher scores indicating worse outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States